CLINICAL TRIAL: NCT02156518
Title: Investigating the Efficacy of Vocal Function Exercises in the Treatment of Voice Problems in Adults Treated With Radiation Therapy for Laryngeal Cancers
Brief Title: The Efficacy of Vocal Function Exercises for Laryngeal Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrushali Angadi (Other)
Responsible Party: Sponsor-Investigator, Vrushali Angadi, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2014-027
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Vocal Folds
Keywords: radiation therapy, laryngeal cancer, voice therapy, vocal function exercises
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vocal Function Exercises (Experimental): Vocal Function Exercises
  Interventions: Procedure: Vocal Function Exercises
- Vocal hygiene (Active Comparator): Vocal hygiene
  Interventions: Procedure: Vocal Hygiene

INTERVENTIONS:
Procedure: Vocal Function Exercises — Vocal Function Exercises
  Arms: Vocal Function Exercises
Procedure: Vocal Hygiene — Vocal Hygiene
  Arms: Vocal hygiene

SUMMARY:
The purpose of this study is to determine if the systematic practice of Vocal Function Exercises (VFE) improves selected measures of voice production in participants who have previously been irradiated for early glottic cancers compared to participants who receive the present standard of care, namely, vocal hygiene counseling. It is hypothesized that a prescriptive vocal exercise program (VFE) will improve the voice production of individuals who have been previously treated for laryngeal cancers when compared to participants who receive vocal hygiene alone.

ELIGIBILITY:
Inclusion Criteria:

* Hearing level and cognitive ability to follow test directions
* Laryngeal cancer
* Radiation Therapy completed >= 6 months
* Deemed disease free by the treating physician
* Subjects have to be willing to attend weekly voice therapy sessions

Exclusion Criteria:

* Adjuvant treatment: laser or any surgical intervention
* Neurological or cognitive impairment
* Hearing levels that interfere with following test instruction
* Vocal fold paralysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Voice production | 6 weeks
  Voice Handicap Index, a validated self- assessment tool was used as the primary outcome measure. A score of 0 indicates no handicap, and a score of 120 indicates complete impairment. Data will be presented as pre and post treatment score (pre and post 6 weeks of therapy).

CONTACTS AND LOCATIONS:
Overall Officials: Vrushali Angadi, Principal Investigator — University of Kentucky, Department of Rehabilitation Sciences
Locations (2):
- United States (2):
  - University of Kentucky, Markey Cancer Center, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky